CLINICAL TRIAL: NCT03084120
Title: Effect of the Maternal Obesity and/or the By-pass on the Growth and the Nutritional Balance of the Child
Acronym: SMOOTHIE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Diagnostic
Other Study IDs: 2016-A01546-45
Record Dates: First submitted 2017-02-20; First posted 2017-03-20 (Actual); Last update posted 2017-11-30 (Actual); Status verified 2017-11

CONDITIONS: Maternal Obesity
MeSH Terms: conditions — Pregnancy in Obesity | interventions — Glycation End Products, Advanced

STUDY DESIGN:
Intervention Model Description: a prospective monocentric study, not therapeutic, and physiopathological
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Gastric bypass surgery (Other): Pregnant women having undergone a Gastric bypass surgery before the pregnancy.
  * Collection of bloods samples for the mother.
  * Retrieval of umbilical cord blood.
  * Retrieval of placenta.
  * Collection of newborn's and mother's lock of hair.
  * Dietetic patient outcomes questionnaires for the mother.
  * Parental questionnaires : ASQ (Ages & Stages questionnaires) and CFQ (Child Feeding Questionnaire).
  Interventions: Other: Collection of bloods samples for the mother; Other: Retrieval of umbilical cord blood.; Other: Retrieval of placenta.; Other: Collection of newborn's and mother's lock of hair.; Other: Dietetic Patient Outcomes Questionnaires for the mother.; Other: Parental questionnaires : ASQ (Ages & Stages questionnaires) and CFQ (Child Feeding Questionnaire).
- Reference group (Other): Pregnant women having a body mass index <25 kg/m2 at the early pregnancy.
  * Collection of bloods samples for the mother.
  * Retrieval of umbilical cord blood.
  * Retrieval of placenta.
  * Collection of newborn's and mother's lock of hair.
  * Dietetic patient outcomes questionnaires for the mother.
  * Parental questionnaires : ASQ (Ages & Stages questionnaires) and CFQ (Child Feeding Questionnaire).
  Interventions: Other: Collection of bloods samples for the mother; Other: Retrieval of umbilical cord blood.; Other: Retrieval of placenta.; Other: Collection of newborn's and mother's lock of hair.; Other: Dietetic Patient Outcomes Questionnaires for the mother.; Other: Parental questionnaires : ASQ (Ages & Stages questionnaires) and CFQ (Child Feeding Questionnaire).
- Overweight (Other): Pregnant women having a body mass index 25-30 kg/m2 at the early pregnancy.
  * Collection of bloods samples for the mother.
  * Retrieval of umbilical cord blood.
  * Retrieval of placenta.
  * Collection of newborn's and mother's lock of hair.
  * Dietetic patient outcomes questionnaires for the mother.
  * Parental questionnaires : ASQ (Ages & Stages questionnaires) and CFQ (Child Feeding Questionnaire).
  Interventions: Other: Collection of bloods samples for the mother; Other: Retrieval of umbilical cord blood.; Other: Retrieval of placenta.; Other: Collection of newborn's and mother's lock of hair.; Other: Dietetic Patient Outcomes Questionnaires for the mother.; Other: Parental questionnaires : ASQ (Ages & Stages questionnaires) and CFQ (Child Feeding Questionnaire).
- Obesity (Other): Pregnant women having a body mass index > 30 kg/m2 at the early pregnancy.
  * Collection of bloods samples for the mother.
  * Retrieval of umbilical cord blood.
  * Retrieval of placenta.
  * Collection of newborn's and mother's lock of hair.
  * Dietetic patient outcomes questionnaires for the mother.
  * Parental questionnaires : ASQ (Ages & Stages questionnaires) and CFQ (Child Feeding Questionnaire).
  Interventions: Other: Collection of bloods samples for the mother; Other: Retrieval of umbilical cord blood.; Other: Retrieval of placenta.; Other: Collection of newborn's and mother's lock of hair.; Other: Dietetic Patient Outcomes Questionnaires for the mother.; Other: Parental questionnaires : ASQ (Ages & Stages questionnaires) and CFQ (Child Feeding Questionnaire).

INTERVENTIONS:
Other: Collection of bloods samples for the mother — -During pregnancy, childbirth and after delivery
Other: Retrieval of umbilical cord blood. — -During childbirth
Other: Retrieval of placenta. — -During childbirth
Other: Collection of newborn's and mother's lock of hair. — -During childbirth
Other: Dietetic Patient Outcomes Questionnaires for the mother. — -During pregnancy and after delivery
Other: Parental questionnaires : ASQ (Ages & Stages questionnaires) and CFQ (Child Feeding Questionnaire). — -At 2 years of age

SUMMARY:
This study evaluates effect of the Maternal Obesity and/or the By-pass on the Growth and the Nutritional Balance of the Child.The data stemming from mothers presenting obesity or an overweight during their pregnancy and the data stemming from mothers having had a by-pass will be compared with the data stemming from mothers with a normal BMI (Body Mass Index), considered as a reference group. It's the same for the data stemming from newborn children. The newborn children stemming from groups of obese mothers or in overweight will be compared with the data stemming from mothers belonging to the reference group.

DETAILED DESCRIPTION:
The obesity represents a major problem of public health, not only in terms of inferred morbi-mortality but also in terms of economic responsibility. More than 50 % of the women old enough to procreate and 25 % of the women pregnant in Europe are in overweights or obese women. This rate does not stop increasing with prevalence which doubled in 30 years. The overweight or the maternal obesity expose the mother and the child to a greater risk of morbi-mortality. The nutritional stress to which is exposed the foetus during the pregnancy can even have long-term effects with a risk increased by overweight or obesity at the grown-up age, so participating in the cycle of the obesity (" Developmental Origins of Behaviour, Health, and Disease " (DOBHaD) concept).

The morbid obesity (IMC > 40 kg / m2) concern 1 to 3 % of the pregnant women. The gastric bypass surgery is envisaged in case of morbid obesity when the other treatments failed, with better results on the loss of weight and on the comorbidity associated with the obesity, in comparison with not surgical interventions. Near half of the patients who resort to the gastric bypass surgery are women old enough to procreate. Recent studies however moderated the beneficial effects of such an intervention with in particular a greater risk of intra-uterine delay of growth and possible nutritional deficiencies on the descent. The neonatal evaluation was limited to the clinical evaluation, and no biological evaluation of the vitamin and nutritional deficiencies on the growth of the foetus and the placenta was brought reported.

The placenta regulates the contribution in nutriments and oxygen and participle in the foetal homéostasie. The reactive placentary adaptations to an environment of surnutrition or the undernutrition can pull modifications of setting-up, development, functions of the placenta with genic modifications and épigénétiques. All these modifications intervene in a "critical window" in terms of development and participate in the phenomena of foetal programming.

Our working hypothesis is that the nutritional stress in utero associated with the maternal obesity and/or with the by-pass has a medium and long-term short-term, metabolic and neurodevelopmental nutritional impact on the descent.

ELIGIBILITY:
Inclusion Criteria:

* For "Gastric Bypass Surgery" arm :

  * Pregnant women having undergone a Gastric bypass surgery before the pregnancy.
* For "Reference group" arm :

  * Pregnant women having a body mass index < 25 kg/m2 at the early pregnancy.
* For "Overweight" arm :

  * Pregnant women having a body mass index 25-30 kg/m2 at the early pregnancy.
* For "Obesity " arm :

  * Pregnant women having a body mass index > 30 kg/m2 at the early pregnancy.

Exclusion Criteria:

* For every arms :

  * Underage women
  * Woman with a multiple pregnancy

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2017-05-10 (Actual); Primary Completion 2022-08-01 (Estimated); Study Completion 2022-08-01 (Estimated)

PRIMARY OUTCOMES:
Born measurement (weight) expressed in z-score. | At the childbirth
  Z-scores are "pure numbers" (have no units of measurement attached to them).
Born measurement (height) expressed in z-score. | At the childbirth
  Z-scores are "pure numbers" (have no units of measurement attached to them).
Born measurement (cranial perimeter) expressed in z-score. | At the childbirth.
  Z-scores are "pure numbers" (have no units of measurement attached to them).

SECONDARY OUTCOMES:
Modification of auxological data (weight) at the age of 2. | At the age of 2.
  Weight expressed in kilograms.
Modification of auxological data (height) at the age of 2. | At the age of 2.
  Height expressed in centimeters.
Modification of auxological data (cranial perimeter) at the age of 2. | At the age of 2.
  Cranial perimeter expressed in centimeters.
Modification of auxological data (BMI (Body Mass Index)) at the age of 2. | At the age of 2.
  BMI (Body Mass Index) expressed in kg/m².
Modification of auxological data (speed of growth expressed) at the age of 2. | At the age of 2.
  Speed of growth expressed in centimeters per year.
Neurodevelopmental modifications at the age of 2. | At the age of 2.
  Parental questionnaire : Ages & Stages Questionnaires (ASQ).
Modifications of eating habits at the age of 2. | At the age of 2.
  Parental questionnaire : Child Feeding Questionnaire (CFQ).
Vitamin dosages and micronutrients in the blood of cordon. | At the childbirth.
  Dosages.
Vitamin dosages and maternal micronutrients in the first, second, third quarter of the pregnancy, at the childbirth and in 2 months after delivery. | First, second, third quarter of the pregnancy, at the childbirth and in 2 months after delivery.
  Dosages.

CONTACTS AND LOCATIONS:
Overall Officials: Geraldine GASCOIN, Pr, Principal Investigator — University Hospital, Angers
Locations (1):
- UHAngers, Angers, France

IPD SHARING:
Plan to Share IPD: No